CLINICAL TRIAL: NCT02710318
Title: Synchronized Immunization NotifiCations
Acronym: SINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York Presbyterian Hospital (Other); Seattle Children's Hospital (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAP6516; 5R01HS023582-03 (AHRQ)
Record Dates: First submitted 2016-03-12; First posted 2016-03-16 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Vaccination
Keywords: Immunizations; Immunization Information System (IIS); Immunization notifications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunization Alert on (Experimental): Children with visits seen when the immunization alert is on
  Interventions: Behavioral: Electronic immunization alert
- Immunization Alert off (No Intervention): Children with visits seen when the alert is off

INTERVENTIONS:
Behavioral: Electronic immunization alert — Immunization alert in the electronic health record
  Arms: Immunization Alert on

SUMMARY:
Immunization is one of the most effective public health interventions. Yet, nationally coverage has consistently fallen short of national goals, and has remained for the most part stagnant. The continued presence of vaccine-preventable diseases poses a threat to public health. In addition to needed improvement of immunization coverage for the general pediatric/adolescent population, some children with chronic medical conditions need specific additional immunizations, yet many fail to receive them.

Immunization reminders for providers in the electronic health record (EHR) are a type of clinical decision support (CDS) that can reduce missed immunization opportunities. One limitation of these reminders is that they generally depend only on data local to the EHR, which can be incomplete due to record scatter, leading to inaccurate alerts. An Immunization Information System (IIS), also known as an immunization registry, is a population-based system that collects immunization data primarily for children and adolescents from providers at a regional or state level.

The investigators seek to couple bidirectional exchange of IIS immunization information and forecasting tools with patient level medical history from the EHR to deliver accurate, patient-specific EHR immunization reminders.

DETAILED DESCRIPTION:
National immunization coverage has consistently fallen short of Healthy People 2010 and 2020 goals and has remained relatively stagnant over the past few years for many immunizations. One important group with a high risk of under-immunization are children with chronic medical conditions (CMCs), who are also at increased risk of serious morbidity and even death from vaccine preventable diseases. One of the key interventions to improve immunization coverage in both the general population and children with CMCs is to decrease missed opportunities for immunization. Immunization reminders in the electronic health record (EHR) are a type of clinical decision support (CDS) that can reduce missed opportunities. In a recent project, the investigators successfully employed such reminders to increase influenza immunization.

One limitation of EHR immunization reminders is that they generally act only on local EHR immunization data. If that data is incomplete, a provider may be erroneously alerted to order an immunization the child does not need. The likelihood of incomplete local data is high. Nearly one-quarter of children in the U.S. visit more than one immunization provider in their first three years of life, leading to fragmented and incomplete records. Low-income and minority children are especially susceptible to immunization record fragmentation as they are more likely to receive care from multiple clinics and providers. Children with CMCs are also at high-risk since their care is often shared between a primary care provider and subspecialists.Harnessing Immunization Information Systems (IIS) data can help overcome this limitation. IIS are population-based systems that collect immunization data primarily for children and adolescents from providers at a regional or state level, consolidating patient's immunization data into a single location no matter where administered. There are currently IIS in 50 states, five cities, and the District of Columbia. However, in most cases, IIS data are available to providers only on the IIS's website. Yet, frontline care providers are most likely to benefit when an IIS provides information at point of patient care within their EHR workflow. This type of bidirectional exchange of immunization information between IIS and EHR systems is a proposed Stage 3 Meaningful Use objective; this consolidated data would be the most complete data to use for an EHR reminder, but is rarely used.

Another challenge associated with EHR-based immunization reminders is that pediatric and adolescent immunization schedules are complex, requiring up to 35 immunizations plus the annual influenza vaccine. Each immunization series has its own minimum age and dosing intervals, and new immunizations are not uncommon. However, many EHRs may not have or aggressively maintain comprehensive immunization decision rules.

IIS can help overcome this limitation as well. Many include tools for forecasting when doses are next due and can provide that information during data exchange with an EHR, but that has not been assessed.

Bringing IIS immunization data and forecasting tools into a local EHR to power CDS will be helpful for the general population. However, one limitation of immunization CDS, whether provided by an IIS or native to the EHR, is that it does not account for subtleties required by children with certain CMCs who may need extra immunizations specific to their condition or cannot receive certain immunizations. A logical next-step is to couple exchange of IIS immunization data and forecasting tools with patient-level EHR information regarding medical conditions to power accurate, patient-specific EHR immunization reminders. This has yet to be done.

Aim 1: Assess the impact of EHR reminders integrated with immunization data and forecasting from a regional IIS on receipt of generally recommended immunizations in a low-income, urban, pediatric and adolescent population.

Aim 2: Assess the impact of integrated EHR reminders that also incorporate patient's medical conditions on receipt of immunizations specifically recommended for children and adolescents with chronic medical conditions.

Hypothesis 1: Lower rates of under-immunization will be observed when reminders are 'on' vs. 'off'.

Hypothesis 2: Lower rates of over-immunization will be observed when reminders are 'on' vs. 'off'.

Hypothesis 3: Higher rates of captured opportunities will be observed when reminders are 'on' vs. 'off'.

Hypothesis 4: There will be no difference in reminder impact on generally recommended immunizations for children with and without chronic medical conditions (CMCs)

In this three-year project, investigators will conduct a randomized cluster crossover pragmatic clinical trial to assess immunization outcomes during periods when an integrated immunization reminder is 'on' vs. 'off' for generally recommended immunizations as well as ones specific for children with CMCs. The proposed work will generate empiric knowledge regarding the best practices for implementing IIS-supported immunization reminders for both children with and without CMCs. The results may help guide local and national efforts on both immunization data exchange and EHR reminders.

ELIGIBILITY:
Inclusion Criteria:

* medical visit at study site during analytic period

Exclusion Criteria:

* none

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15348 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Under-immunization- general recommendations | 1 day
  Percent of children and adolescents seen during the study periods who are overdue for at least one age appropriate immunization as recommended by the CDC's Advisory Committee on Immunization Practices
Under-immunization- recommendations for children with chronic medical conditions | 1 day
  Percent of children and adolescents with a chronic medical condition for which a specific additional immunization is recommended who are seen during the study periods who are overdue for at least one of these specific immunizations
Over-immunization | 1 day
  Percent of children who have received at least one immunization in excess of the recommended immunizations for their age or condition

SECONDARY OUTCOMES:
Captured opportunity | 1 day
  Proportion of medical visits in the analytic period during which a child/adolescent was eligible for an immunization, and received it

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center/ NewYork Presbyterian Hospital Ambulatory Care Network, New York, New York
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephens AB, Wynn CS, Hofstetter AM, Kolff C, Pena O, Kahn E, Dasgupta B, Natarajan K, Vawdrey DK, Lane MM, Robbins-Milne L, Ramakrishnan R, Holleran S, Stockwell MS. Effect of Electronic Health Record Reminders for Routine Immunizations and Immunizations Needed for Chronic Medical Conditions. Appl Clin Inform. 2021 Oct;12(5):1101-1109. doi: 10.1055/s-0041-1739516. Epub 2021 Dec 15. PMID 34911126